CLINICAL TRIAL: NCT05579119
Title: Efficacy and Safety of Sitagliptin and Glargine Compared to a Basal-plus Insulin Regimen in Hospitalized Patients With Type 2 Diabetes
Brief Title: SITAgliptin Plus GLARgine to Glycemic Control in the Hospital Setting (SITAGLAR-H)
Acronym: SITAGLAR-H
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Especialidades, Centro Medico Nacional "La Raza", Instituto Mexicano del Seguro Social (Other)
Collaborators: National Polytechnic Institute, Mexico (Other)
Responsible Party: Principal Investigator, Abraham Edgar Gracia-Ramos, Principal investigator, Centro Medico Nacional La Raza, IMSS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2021-3501-078
Record Dates: First submitted 2022-07-06; First posted 2022-10-13 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin + glargine (Experimental): Sitagliptin and glargine once daily + correction doses of lispro if needed.
  Interventions: Drug: Sitagliptin 100mg; Drug: Glargine; Drug: Lispro
- Basal-plus (Active Comparator): Glargine once daily plus correction doses of lispro if needed.
  Interventions: Drug: Glargine; Drug: Lispro

INTERVENTIONS:
Drug: Sitagliptin 100mg — Sitagliptin 100 mg po once daily.
  Other Names: Januvia
  Arms: Sitagliptin + glargine
Drug: Glargine — Glargine once daily.
  Other Names: Lantus
Drug: Lispro — Correctional doses of lispro if needed for elevated blood glucose using sliding scale insulin (SSI).
  Other Names: Humalog

SUMMARY:
In noncritically hospitalized patients, hyperglycemia (defined as blood glucose [BG] levels >140 mg/dL) is a common, serious, and costly healthcare problem. On the other hand, the treatment of hyperglycemia is associated with decreased mortality and morbidity. Therefore, clinical guidelines from professional organizations recommend using subcutaneous insulin as the preferred therapy in hospitalized patients in a non-intensive care unit setting (target glucose range 100 - 180 mg/dl). The most recommended regimen is basal-bolus insulin therapy, although this regimen requires multiple daily insulin injections and is associated with a significant risk of hypoglycemia (reported in up to 32%). Thus, a more straightforward regimen that results in similar glycemic efficacy to basal-bolus insulin with less risk of hypoglycemia could improve care for this group of patients.

The basal-plus insulin regimen consists of a daily dose of basal insulin with supplemental (corrective) doses of rapid-acting insulin analogue before meals. This has similar efficacy and safety as the basal-bolus regimen. However, the basal-plus scheme does not provide prandial coverage of insulin.

In another vein, dipeptidyl peptidase-4 (DPP-4) inhibitors are a class of oral glucose-lowering agents that reduce the breakdown of endogenous glucagon-like peptide-1 (GLP-1), stimulating insulin secretion in a glucose-dependent manner. Some clinical trials have demonstrated that DPP-4 inhibitors, in combination with insulin, result in similar improvement in glycemic control and lower rates of hypoglycemia compared to basal-bolus insulin regimens.

For the above, using a long-acting insulin analogue with a DPP-4 inhibitor could provide better glycemic control basal and prandial, and this scheme could represent an alternative to using a basal-plus regimen alone.

In the present study, the investigators will conduct a prospective randomized clinical trial (RCT) to compare the DPP-4 inhibitor, sitagliptin, combined with basal-plus insulin therapy and basal-plus insulin scheme alone in non-critical hospitalized patients.

DETAILED DESCRIPTION:
Patients with a known history of diabetes will be randomized to receive sitagliptin plus basal (glargine) insulin or a basal-plus regimen with glargine. Both groups will receive correction doses of rapid-acting insulin lispro in the presence of hyperglycemia (BG >180 mg/dL) per sliding scale. The overall hypothesis is that treatment with sitagliptin in combination with basal insulin will result in better glycemic control and a lower frequency of hypoglycemic events than treatment with a basal-plus insulin regimen in patients with type 2 diabetes in the hospital setting.

68 subjects with type 2 diabetes will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or female medical non-ICU patients aged 18 - 70 years.
2. A known history of type 2 diabetes > 3 months, receiving either diet alone, oral antidiabetic agents (excluding DPP4 inhibitors), or low-dose (≤ 0.5 units/kg/day) insulin therapy.
3. Subjects with BG >180 mg and < 400 mg/dL at the time of randomization without laboratory evidence of diabetic ketoacidosis (serum bicarbonate < 18 mEq/L or positive serum or urinary ketones).
4. Written informed consent.

Exclusion Criteria:

1. Age < 18 or > 70 years.
2. Subjects with increased BG concentration but without a history of diabetes (stress hyperglycemia).
3. Subjects with a history of type 1 diabetes.
4. Patients with a history of diabetic ketoacidosis or hyperosmolar state.
5. Acute critical illness or coronary artery bypass graft (CABG) surgery is expected to require admission to a critical care unit.
6. Subjects with gastrointestinal obstruction, adynamic ileus, or those expected to require gastrointestinal suction.
7. Unable to take oral food or medications.
8. Patients with clinically relevant pancreatic or gallbladder disease.
9. Patients with significant hepatic disease (Child-Pugh score B or C) or impaired renal function (GFR < 50 ml/min).
10. Treatment with oral or injectable corticosteroid.
11. Mental condition renders the subject unable to understand the study's nature, scope, and possible consequences.
12. Female subjects are pregnant or breastfeeding at the time of enrollment into the study.
13. Hypersensitivity to sitagliptin or another contraindication to DPP4 inhibitors.
14. Subject unable to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Change of the mean daily blood glucose levels during hospital | During hospitalization
  Change of the mean daily blood glucose during the hospitalization between the groups

SECONDARY OUTCOMES:
Percentage of blood glucose readings in 100-180 mg/dL range | During hospitalization, up to 10 days
  Percentage of BG readings in the desired range of 100-180 mg/dl out of all avaialble BG readings.
Dose of Insulin | During hospitalization, up to 10 days
  Average daily amount of insulin used.
Incidence of hypoglycemia (BG <70 mg/dL) | During hospitalization, up to 10 days
  Number of BG readings <70 mg/dL in each group.
Percentage of blood glucose reading >180 mg/dL | During hospitalization, up to 10 days
  Percentage of BG reading >180 mg/dL
Mean length of stay in days in the hospital among different groups | During hospitalization, up to 10 days
  The duration of stay in days in the hospital between the two groups is calculated and mean number of days is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Edgar Gracia-Ramos, MD, MSc, Principal Investigator — Hospital General, Centro Médico Nacional "La Raza", IMSS
Locations (1):
- División de Investigación en Salud, Hospital de Especialidades, Centro Médico Nacional "La Raza", IMSS, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gracia-Ramos AE. Role of incretin-based therapy in hospitalized patients with type 2 diabetes. J Diabetes Investig. 2020 Mar;11(2):508-509. doi: 10.1111/jdi.13130. Epub 2019 Sep 17. PMID 31529777
- [Background] Gracia-Ramos AE, Carretero-Gomez J, Mendez CE, Carrasco-Sanchez FJ. Evidence-based therapeutics for hyperglycemia in hospitalized noncritically ill patients. Curr Med Res Opin. 2022 Jan;38(1):43-53. doi: 10.1080/03007995.2021.1997288. Epub 2021 Nov 22. PMID 34694181
- [Background] Gracia-Ramos AE, Cruz-Dominguez MP, Madrigal-Santillan EO. Incretin-based therapy for glycemic control of hospitalized patients with type 2 diabetes: a systematic review. Rev Clin Esp (Barc). 2022 Mar;222(3):180-189. doi: 10.1016/j.rceng.2021.09.003. Epub 2021 Dec 4. PMID 34872879
- [Background] Umpierrez GE, Gianchandani R, Smiley D, Jacobs S, Wesorick DH, Newton C, Farrokhi F, Peng L, Reyes D, Lathkar-Pradhan S, Pasquel F. Safety and efficacy of sitagliptin therapy for the inpatient management of general medicine and surgery patients with type 2 diabetes: a pilot, randomized, controlled study. Diabetes Care. 2013 Nov;36(11):3430-5. doi: 10.2337/dc13-0277. Epub 2013 Jul 22. PMID 23877988
- [Background] Pasquel FJ, Gianchandani R, Rubin DJ, Dungan KM, Anzola I, Gomez PC, Peng L, Hodish I, Bodnar T, Wesorick D, Balakrishnan V, Osei K, Umpierrez GE. Efficacy of sitagliptin for the hospital management of general medicine and surgery patients with type 2 diabetes (Sita-Hospital): a multicentre, prospective, open-label, non-inferiority randomised trial. Lancet Diabetes Endocrinol. 2017 Feb;5(2):125-133. doi: 10.1016/S2213-8587(16)30402-8. Epub 2016 Dec 8. PMID 27964837
- [Background] Vellanki P, Rasouli N, Baldwin D, Alexanian S, Anzola I, Urrutia M, Cardona S, Peng L, Pasquel FJ, Umpierrez GE; Linagliptin Inpatient Research Group. Glycaemic efficacy and safety of linagliptin compared to a basal-bolus insulin regimen in patients with type 2 diabetes undergoing non-cardiac surgery: A multicentre randomized clinical trial. Diabetes Obes Metab. 2019 Apr;21(4):837-843. doi: 10.1111/dom.13587. Epub 2018 Dec 17. PMID 30456796
- [Background] Garg R, Schuman B, Hurwitz S, Metzger C, Bhandari S. Safety and efficacy of saxagliptin for glycemic control in non-critically ill hospitalized patients. BMJ Open Diabetes Res Care. 2017 Mar 29;5(1):e000394. doi: 10.1136/bmjdrc-2017-000394. eCollection 2017. PMID 28405346
- [Background] Guardado-Mendoza R, Garcia-Magana MA, Martinez-Navarro LJ, Macias-Cervantes HE, Aguilar-Guerrero R, Suarez-Perez EL, Aguilar-Garcia A. Effect of linagliptin plus insulin in comparison to insulin alone on metabolic control and prognosis in hospitalized patients with SARS-CoV-2 infection. Sci Rep. 2022 Jan 11;12(1):536. doi: 10.1038/s41598-021-04511-1. PMID 35017617
- [Derived] Gracia-Ramos AE, Cruz-Dominguez MDP, Madrigal-Santillan EO, Rojas-Martinez R, Morales-Gonzalez JA, Morales-Gonzalez A, Hernandez-Espinoza M, Vargas-Penafiel J, Tapia-Gonzalez MLA. Efficacy and safety of sitagliptin with basal-plus insulin regimen versus insulin alone in non-critically ill hospitalized patients with type 2 diabetes: SITA-PLUS hospital trial. J Diabetes Complications. 2024 May;38(5):108742. doi: 10.1016/j.jdiacomp.2024.108742. Epub 2024 Apr 3. PMID 38581842